CLINICAL TRIAL: NCT01474187
Title: Genotype-driven Phase I Study of Irinotecan Administered in Neoadjuvant Chemoradiotherapy in Patients With Stage II/III Rectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhu Ji, Chief of Department of Radiation Oncology, Cancer Hospital, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-003
Record Dates: First submitted 2011-11-11; First posted 2011-11-18 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Rectal Cancer
Keywords: Neoadjuvant chemotherapy; rectal cancer; phase I study; irinotecan
MeSH Terms: conditions — Rectal Neoplasms | interventions — Irinotecan; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan (Experimental): irinotecan dose initial from 50mg/m2/week, increased by 15mg/mg/week
  Interventions: Drug: Irinotecan; Drug: Capecitabine; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Irinotecan — initial from 50mg/m2/week and increased by 15mg/m2/week
Drug: Capecitabine — 625mg/m2,bid,d1-5,qw
  Other Names: Xeloda
Radiation: Radiotherapy — 50Gy for whole pelvis

SUMMARY:
Irinotecan is one of effective drugs for colorectal cancer. In neoadjuvant chemoradiotherapy (CRT), Irinotecan is prescribed in a low dose of 50mg/m2/week because of toxicity. Some current studies showed that irinotecan's dose can be increased significantly for those patients with 6/6 or 6/7 genotype of UGT1A1. therefore, the investigators designed this trial to explore the maximal tolerable dose (MTD) of Irinotecan in combined neoadjuvant CRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal adenocarcinoma
* Clinical staged T3/4 or any node-positive disease
* Age of 18-75 years
* Karnofsky Performance Status > 80
* Adequate bone marrow reserve, renal and hepatic functions
* Without previous antitumoural chemotherapy
* No evidence of metastatic disease
* Written informed consent before randomization
* UGT1A1's genotype of 6/6 or 6/7

Exclusion Criteria:

* Clinical staged I or IV
* Age of <18 or >75 years
* Karnofsky Performance Status < 80
* Previous pelvis radiotherapy
* Previous antitumoural chemotherapy
* Clinically significant internal disease
* Refuse to write informed consent before randomization
* UGT1A1's genotype of 7/7

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
toxicity | 5 weeks
  * Grade 4 hemato-toxicity
  * Grade 3 nonhemato-toxicity (not include grade 3 anal verge skin toxicity)

SECONDARY OUTCOMES:
pathological complete response (pCR) | within 14days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality, China